CLINICAL TRIAL: NCT00044122
Title: Regulation of the Proliferation and Survival of Normal and Neoplastic Human Mast Cells
Brief Title: Study of Factors Regulating Mast Cell Proliferation
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020277; 02-I-0277
Record Dates: First submitted 2002-08-17; First posted 2002-08-19 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-08-29

CONDITIONS: Mastocytosis; Monoclonal; Bone Marrow; Tryptase
Keywords: Mastocytosis; Natural History
MeSH Terms: conditions — Mastocytosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Adult Relatives: Relatives of patient with mastocytosis
- Adults with Mastocytosis: Adults with documented mastocytosis
- Pediatric Patients with Mastocytosis: Pediatric patients with documented mastocytosis
- Pediatric Relatives: Pediatric relatives of patients with mastocytosis

SUMMARY:
This study will examine growth factors that promote and inhibit mast cell proliferation resulting in mastocytosis, a disease of excessive mast cells in the body. These cells can release chemicals that cause itching, blisters, flushing, bone pain and abdominal pain.

Patients up to 80 years of age with mastocytosis may be eligible for this 1-day study. Participants will have one visit at NIH lasting up to 8 hours, during which they will undergo the following tests and procedures:

* Medical history and physical examination.
* Laboratory studies, if medically indicated.
* Blood tests to identify genetic changes important in the growth, development, and functioning of mast cells.
* Bone marrow aspiration and biopsy.

For the bone marrow procedure, the skin over the hipbone and the outer surface of the bone itself are numbed with local anesthesia. Then, a special needle is inserted into the hipbone and about 1 tablespoon of bone marrow is drawn into a syringe. Another needle is inserted into the same area to collect a small piece of the bone marrow. Additional procedures may include allergen testing, urinalysis, and 24-hour urine collection.

Participants will receive an evaluation of their mastocytosis.

...

DETAILED DESCRIPTION:
This protocol is designed to examine those growth potentiating and inhibiting factors which regulate mast cell number and survival in patients with mastocytosis, and to explore the molecular basis of the disease process in hopes of improving therapy. Patients will carry the diagnosis of mastocytosis based on abnormal bone marrow biopsy and aspirate, abnormal skin biopsy, presence of urticaria pigmentosa, and if available, elevated serum tryptase level > 20 ng/ml and the presence of aberrant mast cell morphology and surface markers of CD2 and CD25. Mastocytosis patients will include children and adults from zero years to 80 years of age. Unaffected relatives (age 2 to 80 years) may also be enrolled. The protocol is designated for up to a 1-year enrollment period; with only a small number of enrolled patients that will stay on study for more than one visit, based on investigator assessment of contribution to study objectives. Participants will undergo standard physical exam, medical history review, and blood collection for clinical and research laboratory evaluations. We will collect clinical data and biological specimens for research evaluation from individuals undergoing clinically indicated diagnostic procedures. Some patients may participate in research evaluations including buccal swab collection, dietary intake assessment, stool collection, exercise challenge, microbiome studies, and activity tracking. These studies are optional. Patients may be asked to re-enter this protocol at a later time for further follow-up.

ELIGIBILITY:
* PATIENT PARTICIPANT INCLUSION CRITERIA:

Participants with mastocytosis zero to 80 years of age may participate in telehealth visits, and two to 80 years of age may participate on-site at NIH Clinical Center.

Histologic evidence of increased mast cell number by bone marrow and/or skin biopsy or documentation of mastocytosis in the skin

supported with a photograph of diagnostic skin lesions

Must be under the care of a primary care physician to be enrolled.

Ability to provide informed consent.

PATIENT PARTICIPANT EXCLUSION CRITERIA:

Anemia with hemoglobin less than 8 g/dL, hematocrit less than 24.

Any condition that in the opinion of the investigator contraindicates participation in this study.

RELATIVE INCLUSION CRITERIA:

Two to 80 years of age.

A biological relative without the diagnosis of mastocytosis by skin examination or histologic evidence in a skin or bone marrow biopsy

Participant has a primary medical care provider outside the NIH

Ability to provide informed consent.

RELATIVE EXCLUSION CRITERIA:

Any condition that in the opinion of the investigator contraindicates participation in this study.

Ages: 1 Day to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: primary clinical
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2002-09-18 (Actual)

PRIMARY OUTCOMES:
To obtain normal and neoplastic human mast cells from the bone marrow and peripheral blood of patients with mastocytosis in order to study the regulation of the proliferation and survival of these cells, and to assess the extent and classificati... | Patients return to NIH as necessary
  continuing collection of cells from subjects with mastocytosis for ongoing experimentation in laboratory

CONTACTS AND LOCATIONS:
Overall Officials: Hirsh D Komarow, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carter MC, Metcalfe DD, Komarow HD. Mastocytosis. Immunol Allergy Clin North Am. 2014 Feb;34(1):181-96. doi: 10.1016/j.iac.2013.09.001. Epub 2013 Oct 7. PMID 24262698
- [Background] Chan EC, Bai Y, Kirshenbaum AS, Fischer ER, Simakova O, Bandara G, Scott LM, Wisch LB, Cantave D, Carter MC, Lewis JC, Noel P, Maric I, Gilfillan AM, Metcalfe DD, Wilson TM. Mastocytosis associated with a rare germline KIT K509I mutation displays a well-differentiated mast cell phenotype. J Allergy Clin Immunol. 2014 Jul;134(1):178-87. doi: 10.1016/j.jaci.2013.12.1090. Epub 2014 Feb 28. PMID 24582309
- [Background] Cruse G, Metcalfe DD, Olivera A. Functional deregulation of KIT: link to mast cell proliferative diseases and other neoplasms. Immunol Allergy Clin North Am. 2014 May;34(2):219-37. doi: 10.1016/j.iac.2014.01.002. Epub 2014 Mar 12. PMID 24745671
- [Derived] Krausfeldt LE, Cao V, Rodrigues R, Henderson WA, Eisch R, Scott LM, Metcalfe DD, Komarow HD. Evidence for dysbiosis in the gut microbiome of patients with systemic mastocytosis. J Allergy Clin Immunol Glob. 2025 Oct 9;5(1):100578. doi: 10.1016/j.jacig.2025.100578. eCollection 2026 Jan. PMID 41583012
- [Derived] Wilson TM, Maric I, Simakova O, Bai Y, Chan EC, Olivares N, Carter M, Maric D, Robyn J, Metcalfe DD. Clonal analysis of NRAS activating mutations in KIT-D816V systemic mastocytosis. Haematologica. 2011 Mar;96(3):459-63. doi: 10.3324/haematol.2010.031690. Epub 2010 Dec 6. PMID 21134978
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2002-I-0277.html